CLINICAL TRIAL: NCT03099343
Title: Location-based Tailored Messaging to Reduce Sodium Intake in Hypertensive Patients
Brief Title: Tailored Messaging to Reduce Sodium Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott L. Hummel, MD MS Assistant Professor Internal Medicine Cardiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00123069
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
Keywords: sodium; salt; diet; tailored messaging; mobile application
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Location-based Tailored Messaging (Experimental): Participants receive location-based tailored messaging via a mobile application throughout the 8-week research study.
  Interventions: Behavioral: Location-based Tailored Messaging
- Control Group (No Intervention): Participants follow their usual eating pattern and will not have access to the application throughout the 8-week research study.

INTERVENTIONS:
Behavioral: Location-based Tailored Messaging — The mobile application works by providing tailored messages targeted to participant locations that can help individuals to choose lower sodium foods.
  Arms: Location-based Tailored Messaging

SUMMARY:
The proposed study will determine the effectiveness of a mobile application location-based tailored notification message system in helping hypertensive patients reduce dietary sodium intake and feel more confident in following a low sodium diet.

DETAILED DESCRIPTION:
People with high blood pressure often get advice to lower their salt or sodium intake. High dietary sodium intake is linked to high blood pressure, stroke, heart failure and kidney disease. U.S. federal guidelines advocate daily sodium intake of less than 2,300 milligrams (mg). The estimated average sodium intake for Americans is 3,400 mg per day. In recent years, consumption of processed and restaurant foods has substantially increased. More than 75% of sodium in the average U.S. diet now comes from these sources.

The mobile application will deliver tailored messages based on the user's location and previously identified high-sodium food items that they commonly consume.

This 8-week research study at Visit 1 or baseline will consent and randomize 50 eligible adults with high blood pressure to use the mobile application daily or to follow their usual eating pattern with no access to the application.

All participants will be asked to complete four surveys at baseline and Week 8: Block Food Frequency Questionnaire, Block Sodium Screener, Self-care Confidence in following a Low Sodium Diet and the Automated Self-administered 24-Hour Dietary Recall survey. All participants will be asked to provide a baseline and end of study 24-hour urine collection, regularly provide home blood pressure measurements and urine dipstick tests every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Hypertension
* Use of anti-hypertensive therapy for at least 3 months, with stable anti-hypertensive therapy (medication type and dose) for at least 2 weeks
* Daily sodium intake of >2,000 mg with sodium to kcal ratio > 1, estimated via Food Frequency Questionnaire
* Ownership and use of an Apple iPhone

Exclusion Criteria:

* Chronic Kidney Disease
* Heart Failure
* Systolic Blood Pressure >180 mm Hg
* Diastolic Blood Pressure >110 mm Hg
* Use of a loop diuretic or corticosteroid
* Insulin dependent diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
24-hour urinary sodium excretion | Baseline, Week 8
  Change from baseline in 24-hour urinary sodium excretion at week 8
Self-care Confidence in Following a Low-sodium Diet Scale (SCFLDS) | Baseline, Week 8
  Change from baseline in Self-care Confidence in Following a Low-sodium Diet Scale (SCFLDS) at week 8. It assesses the participants' confidence in the ability to select and prepare low-sodium foods. The self-reported tool consists of 7 items with 4 response options per item. The score range is 1-4 (1=Not confident, 2=Somewhat confident, 3=Very confident, 4=Extremely confident) then added for each question. Possible scores range from 7 to 28 and the higher the score indicates greater confidence.

OTHER OUTCOMES:
Change from baseline in blood pressure | Baseline, week 8
  Change in home-measured brachial cuff blood pressure
Estimated dietary sodium intake | Baseline, week 8
  Estimated dietary sodium intake from Block Food Frequency Questionnaire (inter-group comparison at week 8, intra-group change from baseline-week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Hummel, MD, MS, Principal Investigator — University of Michigan; Michael P Dorsch, PharmD, MS, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alhashimi L, Cordwin DJ, Dandu C, Hummel SL, Dorsch MP. Patient self-assessment of urine dipsticks to estimate sodium intake in patients with hypertension. Clin Nutr ESPEN. 2022 Oct;51:295-300. doi: 10.1016/j.clnesp.2022.08.011. Epub 2022 Aug 12. PMID 36184219
- [Derived] Dorsch MP, Cornellier ML, Poggi AD, Bilgen F, Chen P, Wu C, An LC, Hummel SL. Effects of a Novel Contextual Just-In-Time Mobile App Intervention (LowSalt4Life) on Sodium Intake in Adults With Hypertension: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Aug 10;8(8):e16696. doi: 10.2196/16696. PMID 32663139
- [Derived] Dorsch MP, An LC, Hummel SL. A Novel Just-in-Time Contextual Mobile App Intervention to Reduce Sodium Intake in Hypertension: Protocol and Rationale for a Randomized Controlled Trial (LowSalt4Life Trial). JMIR Res Protoc. 2018 Dec 7;7(12):e11282. doi: 10.2196/11282. PMID 30530462